CLINICAL TRIAL: NCT02400411
Title: The Effects of Margarine and Ham or Vegetable Soup on the on the Glycemic and Insulinemic Responses Elicited by Whole Grain Rye Bread or White Wheat Bread
Brief Title: The Glycemic and Insulinemic Responses Elicited by Meals Containing Whole Grain Rye Bread or White Wheat Bread
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Fazer Group (Industry)
Responsible Party: Principal Investigator, Mikael Fogelholm, professor, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HY_RAV_Breadmeal
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Blood Glucose Concentration
Keywords: Carbohydrate; Glycemic response; insulin; whole grain; meal
MeSH Terms: conditions — Insulin Resistance | interventions — Margarine; ATF7IP protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Wheat bread (Experimental): Bread-based meal
  Interventions: Other: Wheat bread
- Wheat bread with margarine and ham (Experimental): Bread-based meal
  Interventions: Other: Wheat bread; Other: margarine; Other: ham
- Wheat bread with margarine, ham and soup (Experimental): Bread-based meal
  Interventions: Other: Wheat bread; Other: margarine; Other: ham; Other: soup
- Rye bread (Experimental): Bread-based meal
  Interventions: Other: rye bread
- Rye bread with margarine and ham (Experimental): Bread-based meal
  Interventions: Other: margarine; Other: ham; Other: rye bread
- Rye bread with margarine, ham and soup (Experimental): Bread-based meal
  Interventions: Other: margarine; Other: ham; Other: soup; Other: rye bread

INTERVENTIONS:
Other: Wheat bread
  Arms: Wheat bread; Wheat bread with margarine and ham; Wheat bread with margarine, ham and soup
Other: margarine
  Arms: Rye bread with margarine and ham; Rye bread with margarine, ham and soup; Wheat bread with margarine and ham; Wheat bread with margarine, ham and soup
Other: ham
  Arms: Rye bread with margarine and ham; Rye bread with margarine, ham and soup; Wheat bread with margarine and ham; Wheat bread with margarine, ham and soup
Other: soup
  Arms: Rye bread with margarine, ham and soup; Wheat bread with margarine, ham and soup
Other: rye bread
  Arms: Rye bread; Rye bread with margarine and ham; Rye bread with margarine, ham and soup

SUMMARY:
This is a postprandial study with healthy volunteers. The glycemic and insulinemic responses elicited by meals containing either whole grain rye bread or white wheat bread as such or combined with margarine and ham and vegetable soup are compared. Blood glucose concentrations are monitored from finger prick blood samples collected before the meal and at 15, 30, 45, 60, 90 and 120 min. Venous samples for insulin concentrations are taken at time-points 0, 30 and 60 min.

ELIGIBILITY:
Inclusion Criteria:

* female
* BMI 18-27 kg/m2

Exclusion Criteria:

* pregnant or breastfeeding
* diabetes, gastrointestinal disease
* regular use of medication
* strict vegetarian or vegan diet
* food allergy
* recent blood donation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Blood glucose concentration | 120 min

SECONDARY OUTCOMES:
Serum insulin concentration | 60 min